CLINICAL TRIAL: NCT05187806
Title: Effects of Motivational Interviewing Intervention on Self- Management and HbA1c in Type 2 Diabetes Patients
Brief Title: Motivational Interviewing With Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Deniz KAYA MERAL, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NursePsychiatric
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; motivational interviewing; HbA1c; self management
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Masking Description: Without knowing that participants are in the experimental or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): After the pretest, the experimental group was intervened with a motivational interview (MI) method that consisted of four sessions of 30-60 (mean 45 min) min each. The sessions were structured according to the Behavior Change Stage Identification Form developed by the researcher by making use of the trans-theoretical model and adapting it to diabetic patients. The subject of the first session was "Opening, Structuring the Discussion, and Establishing the Agenda"; the subject of the second session was "Improving Motivation for Change"; the subject of the third session was "Summarizing, Support, and Talking about the Change"; and the subject of the fourth session was "Evaluation" . The discussions were completed in four weeks, with one discussion held every week. The final test and the Diabetes Self-Management Instrument were applied again to the members of the intervention group in the third month after completion of the MI method sessions.
  Interventions: Behavioral: motivational interview
- Control group (No Intervention): The control group received routine treatment. The final test and the Diabetes Self-Management Instrument were applied again to the members of the control group in the third month.

INTERVENTIONS:
Behavioral: motivational interview — After the pretest, the experimental group was intervened with a motivational interview (MI) method that consisted of four sessions.The pretest and posttest Diabetes Self-Management Scale total scores and HbA1c values of the patients in the experimental and control groups were compared.
  Arms: Experimental group

SUMMARY:
This study was conducted in a quasi-experimental research design with a pretest-posttest control group to determine the effect of motivational interviewing on self-management and HbA1c in patients with type 2 diabetes. The sample of the study consisted of 25 experimental and 26 controls, who applied to an outpatient clinic in a training and research hospital.

DETAILED DESCRIPTION:
This study was conducted in a quasi-experimental research design with a pretest-posttest control group to determine the effect of motivational interviewing on self-management and HbA1c in patients with type 2 diabetes. The sample of the study consisted of 25 experimental and 26 controls, who applied to an outpatient clinic in a training and research hospital. After the pretest, the experimental group was intervened with a motivational interview (MI) method that consisted of four sessions; the control group received routine treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Having been diagnosed with type 2 diabetes for more than 3 months
* Being in the contemplation
* Preparation, and/or action stages of any section of the Behavioral Change Stage Identification Form of the Trans-Theoretical Model
* Having HbA1c levels above 6
* Agreeing to take part in the study

Exclusion Criteria:

* Having a perception disorder that will prevent communication
* Having been diagnosed with any mental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years and older
Enrollment: 60 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Comparison of the pretest-posttest Diabetes Self-management Instrument-35 scores | 3 months
  The instrument is comprised of 35 questions covering the period from the previous three months to determine the frequency of the implementation of the self-management skills of the patients. The total score for the Instrument ranged from 35 to 140. A higher score showed that self-management activities were implemented on a more regular basis. Interventions consisted of four sessions of 30-60 (mean 45 min) min each. The sessions were structured according to the Behavior Change Stage Identification Form developed by the researcher by making use of the trans-theoretical model and adapting it to diabetic patients.The discussions were completed in four weeks, with one discussion held every week. The final test and the Diabetes Self-Management Instrument were applied again to the members of the intervention group in the third month after completion of the MI method sessions and in the third month to the control group.

SECONDARY OUTCOMES:
Comparison of the pretest-posttest HbA1c values | 3 months
  The pretest and posttest HbA1c values of the patients in the experimental and control groups were compared in the third month.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Kaya Meral, Phd, Principal Investigator — Ministry of Health, Gaziosmanpasa Training and Research Hospital
Locations (1):
- Ministry of Health, Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share to Individual participant data

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT05187806/Prot_SAP_000.pdf